CLINICAL TRIAL: NCT01514513
Title: A Comparative Study to Demonstrate the Efficacy and Safety of Licefreee Spray Against Nix 1% Permethrin in Head Lice Infested Individuals
Brief Title: Efficacy and Safety of Licefreee Spray Against Nix 1% Permethrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Florida Family Health and Research Centers (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LF001-0011
Record Dates: First submitted 2012-01-11; First posted 2012-01-23 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Pediculosis Capitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Licefreee Spray (Experimental)
  Interventions: Drug: Licefreee Spray
- Nix Creme Rinse, 1% Permethrin (Active Comparator)
  Interventions: Drug: 1% permethrin creme rinse

INTERVENTIONS:
Drug: Licefreee Spray — Liquid applied to hair and left on for at least one hour once on day 1 and once on day 8 if live lice are present.
  Arms: Licefreee Spray
Drug: 1% permethrin creme rinse — Creme rinse applied to hair and rinsed off after 10 minutes once on day 1 and once on day 8 if live lice are present.
  Arms: Nix Creme Rinse, 1% Permethrin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Licefreee Spray in eradicating head lice as compared to Nix, both are available over-the-counter lice treatments.

DETAILED DESCRIPTION:
Head lice is a worldwide problem. Many treatments for lice appear to be losing their effectiveness; therefore products are needed that safely and effectively eradicate lice.

ELIGIBILITY:
Inclusion Criteria:

* Must be 4 years of age or older

  * Must have an active head lice infestation of at least 10 lice and viable nits
  * Agree not used any other pediculicides or medicated products during the study
  * Agree not to use a nit comb during the study
  * Must have a single place of residence

Exclusion Criteria:

* Used any form of head lice treatment, prescription, OTC or home remedy for at least four weeks prior to their visit

  * Used topical medication of any kind on the hair for a period of 48 hours prior to visit
  * Individuals receiving systemic, topical drugs or medications which may interfere with the study results
  * Has a history of allergy or hypersensitivity to ragweed or any ingredient in either test products
  * Individuals with any visible skin/scalp condition at the treatment site which, in the opinion of the investigator, will interfere with the evaluation
  * Females who are pregnant or nursing

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Serrano, Principal Investigator — South Florida Family Health and Research Centers
Locations (1):
- Lice Source Services Inc., Plantation, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Licefreee Spray | Nix Creme Rinse, 1% Permethrin
Started | 21 | 21
Completed | 20 | 20
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Licefreee Spray | Nix Creme Rinse, 1% Permethrin | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Full Range); unit: years] | 15.57 [6 to 43] | 14.76 [4 to 42] | 15.17 [4 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 20 | 33
  Not Hispanic or Latino | 8 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42
Hair Length [Number; unit: participants]
  Extra long | 5 | 3 | 8
  Long | 7 | 6 | 13
  Medium | 7 | 11 | 18
  Short | 2 | 1 | 3
Hair Texture [Number; unit: participants]
  Fine | 8 | 4 | 12
  Average | 10 | 10 | 20
  Coarse | 3 | 7 | 10
Hair Curliness [Number; unit: participants]
  Curly | 1 | 5 | 6
  Wavy | 10 | 8 | 18
  Straight | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: The Proportion Within Each Treatment Group of Subjects Who Have no Live Lice
Description: No live lice 15 days following initial treatment
Time Frame: 15 days
Measure: Number; unit: participants
Arm/Group | Licefreee Spray | Nix Creme Rinse, 1% Permethrin
Number analyzed (Participants) | 20 | 20
participants | 17 | 9

2. Secondary Outcome: Adverse Events
Description: Number of participants with adverse events
Time Frame: 15 days
Measure: Number; unit: participants
Arm/Group | Licefreee Spray | Nix Creme Rinse, 1% Permethrin
Number analyzed (Participants) | 20 | 20
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Licefreee Spray | Nix Creme Rinse, 1% Permethrin
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No